CLINICAL TRIAL: NCT01692730
Title: Web Assisted Tobacco Intervention With Community Colleges
Acronym: WATI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Library of Medicine (NLM) (NIH)
Responsible Party: Principal Investigator, Scott McIntosh, Associate Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RSRB00040730; R01CA152093 (NIH); R01CA152093-01A1 (NIH)
Record Dates: First submitted 2012-09-17; First posted 2012-09-25 (Estimated); Results first posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Tobacco Dependence
Keywords: Smoking Cessation; Web Assisted Tobacco Intervention
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced Web Assisted Intervention (Experimental): Enhanced Web Assisted Tobacco Intervention. An enhanced and highly interactive website for cessation.
  Interventions: Behavioral: Enhanced Web Assisted Tobacco Intervention
- Basic Web Assisted Intervention. (Active Comparator): Basic Web Assisted Tobacco Intervention. A basic website for cessation comparable to those for general adult populations, including established evidence-based cessation information and features.
  Interventions: Behavioral: Basic Web Assisted Tobacco Intervention

INTERVENTIONS:
Behavioral: Enhanced Web Assisted Tobacco Intervention — Subjects at community college campuses will be directed to a cessation website with current Public Health Service Guideline information and effective smoking cessation strategies, and some combination of novel interactive and social network features, including a variety of better-practice features recommended recent literature, and technologically advanced proactive features (e-mails, SMS texting, and social networking).
  Other Names: Smoking Cessation Intervention; Web based smoking cessation
  Arms: Enhanced Web Assisted Intervention
Behavioral: Basic Web Assisted Tobacco Intervention — Subjects at community college campuses will be directed to a cessation website with current Public Health Service Guideline information and effective smoking cessation strategies, and with minimal interactive web-based features.
  Other Names: Static Web Assisted Tobacco Intervention; Information only
  Arms: Basic Web Assisted Intervention.

SUMMARY:
This trial will test the effectiveness of an enhanced web-based smoking cessation intervention for student smokers at 2-year Community Colleges. Young adults continue to be understudied, so more studies of cessation interventions are needed to generate an acceptable level of strength of evidence regarding quit rates, particularly so for Community College students for whom little data on cessation are available. Students (research subjects) will be directed to one of two intervention websites with various levels of novel interactive and social network features, including a variety of better-practice features recommended by recent literature, and technologically advanced proactive features (e-mails, SMS texting, and social networking).

Our study hypothesizes that students with access to an enhanced website will have higher rates of self-reported intention to quit, a higher number of quit attempts at 6-months compared to those in in a non-enhanced website. Overall, this study will evaluate evidence for a novel enhanced cessation intervention model and will add to our understanding of successful intervention with an understudied population of primarily young adult Community College smokers. The intervention components will be replicable and, if effective, the methodology is applicable across populations, and has the potential for broad public health impact through improved delivery of effective stop smoking interventions via the internet.

DETAILED DESCRIPTION:
Purpose of the study. This group randomized controlled trial will test the effectiveness of an enhanced web-based cessation intervention for student smokers at 2-year Community Colleges (CC). Compared to the smoking rates of the general population (18%), smoking rates among CC students varies but remains substantially higher (28-30%). Evaluations of Web-Assisted Tobacco Interventions (WATI) for smoking cessation treatment with young adults in more traditional 4-year college settings have yielded encouraging preliminary data regarding intervention effectiveness. Young adults continue to be understudied, so additional randomized designed studies of cessation interventions are needed to generate an acceptable level of strength of evidence regarding quit rates, particularly so for CC students for whom little data on cessation are available. This critical population is likely to be increasing for several reasons, including President Obama's American Graduation Initiative, which provides resources to increase Community College enrollment by 5 million additional graduates by 2020. In the proposed trial, subjects on campuses randomized to the basic intervention arm will be directed to a minimally interactive website standardized to comply with 2008 DHHS Clinical Practice Guidelines for adult smokers. Those at campuses in the enhanced intervention arm will be directed to an enhanced site that adds novel interactive and social network features, including a variety of better-practice features recommended by WATI workshops, recent literature, and technologically advanced proactive features (e-mails, SMS texting, and social networking). Our study has the following Specific Aims:

Primary Aims Aim 1:To test the effectiveness of an Enhanced interactive WATI (E-WATI) vs. a Basic WATI (B-WATI) among Community College students (primarily young adults). The online methodology will maximize population access and, if effective, can be recommended as a feasible cessation option.

Aim 2:To evaluate both WATI options for overall usability, as well as for the usability and perceived helpfulness of key features (i.e., basic, novel, high-tech, proactive and interactive components), and their relationship to cessation.

Secondary Aim Aim 3:To develop and evaluate strategies to recruit and retain an understudied population of Community College smokers using WATI interventions. Evaluation of recruitment strategies will be useful to the current trial, as well as well as to future trials with this population.

This study will be conducted in three phases, using a mixed methods approach. Phase 1 qualitative research in Year 01 will help guide and refine recruitment and retention and delivery strategies. In Phase 2, a group randomized trial in Years 02-04 will randomize 16 Community Colleges (8 matched pairs; 1,440 smokers) to one of two interventions: 1) B-WATI - a basic website for cessation comparable to those for general adult populations, including established evidence-based cessation information and features; or 2) E-WATI - an enhanced and highly interactive website for cessation. Phase 3 dissemination in Year 05 will involve interpretation of study results, guidance for further research, and dissemination of study findings, including recommendations for including WATI cessation for campus-based referral strategies. To address the Specific Aims, our study has these Primary Hypotheses:

H1.0: Smokers in E-WATI will have higher biochemically verified point-prevalence abstinence at 6-months compared to those in the B-WATI group. Secondary hypotheses for smoking-related outcomes explore: (H1.1) higher rates of self-reported intention to quit; (H1.2), a higher number of quit attempts at 6-months in the E-WATI group compared to those in B-WATI and higher quit rates at 12 months for the subsample available for follow-up; (H1.3) higher number of prolonged abstinence participants at 6-months, and (H1.4), greater movement through Stages of Change.

H2.0: Smokers in the E-WATI group, compared to those in B-WATI, will demonstrate more interactivity and engagement with web-based features and interventions as measured by website usability analysis and higher self-report of the number and type of selected online strategies at 6-month follow-up.

H3.0: Web-based features will be perceived as more helpful for smoking cessation by those in E-WATI compared to those in B-WATI as measured by the 6-month follow-up questionnaire.

Overall, this study will evaluate evidence for a novel enhanced cessation intervention model and will add to our understanding of successful intervention with an understudied population of primarily young adult Community College smokers. The intervention components will be replicable and, if effective, the WATI methodology is applicable across heterogeneous populations and geographic areas, and has the potential for broad public health impact through improved delivery of effective cessation interventions via the internet.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Smoke at least 1 cigarette per day on average
* Attendance at Community College

Exclusion Criteria:

* Age 17 or younger
* Nonsmoker
* Not attending a Community College

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1452 (Actual)
Dates: Start 2012-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott McIntosh, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Derived] McIntosh S, Johnson T, Wall AF, Prokhorov AV, Calabro KS, Ververs D, Assibey-Mensah V, Ossip DJ. Recruitment of Community College Students Into a Web-Assisted Tobacco Intervention Study. JMIR Res Protoc. 2017 May 8;6(5):e79. doi: 10.2196/resprot.6485. PMID 28483741

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Enhanced Web Assisted Intervention | Basic Web Assisted Intervention.
Started | 723 | 729
Completed | 498 | 502
Not Completed | 225 | 227
Not completed — Lost to Follow-up | 225 | 227

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Web Assisted Intervention | Basic Web Assisted Intervention. | Total
Number analyzed (Participants) | 723 | 729 | 1452
Age, Continuous [Mean (Standard Deviation); unit: years] — Collected via online survey.
  years | 27.55048409 (9.474060629) | 28.45541838 (9.707011106) | 28.00482094 (9.602390308)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 26 participants, 11 in EWATI and 15 in BWATI, did not provide sex/gender data.
  Participants
    number analyzed (Participants) | 712 | 714 | 1426
    Female | 237 | 256 | 493
    Male | 475 | 458 | 933

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Self-report Abstinence From Tobacco
Description: Our primary outcome is self-reported abstinence at the six month evaluation point. Abstinence outcomes at this time point are defined in three ways: 1) as self-reported abstinence (no cigarettes or other tobacco use) in the past 7 days prior to this six month time point, 2) or as no use in the past 30 days prior to this six-month time point (the 30 day period is the more conservative measure), or 3) self-reported prolonged abstinence from the time of a specific self-reported cessation date.
Time Frame: 6 month follow-up
Population: The primary outcome time point was six months. These 1,000 participants completed the six month time point evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Web Assisted Intervention | Basic Web Assisted Intervention.
Number analyzed (Participants) | 498 | 502
Participants | 144 | 65

2. Secondary Outcome: Number of Participants With Biochemically Verified Abstinence From Tobacco
Description: Our primary outcome is biochemically-verified point-prevalence abstinence at 6 months. If participant self-reports no cigarettes (or other tobacco use) in the past 7 days, the past 30 days, or since a specific self-reported cessation date, biochemical verification will be conducted to measure salivary cotinine (a cut off of <10ng/ml confirms self-reported abstinence for at least the previous 7 days). Using Intent-to-Treat analysis, subjects who drop out or refuse biochemical verification will be considered smokers.
Time Frame: 6 month follow-up
Population: Not all participants provided saliva. Analysis was performed on a total of 109 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Web Assisted Intervention | Basic Web Assisted Intervention.
Number analyzed (Participants) | 64 | 45
Participants | 35 | 21

ADVERSE EVENTS:
Description: No adverse event data was collected for this study.
Arm/Group | Enhanced Web Assisted Intervention | Basic Web Assisted Intervention.
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes